CLINICAL TRIAL: NCT01465828
Title: PhaRmacodynamic Effects of Switching thErapy in paTients With High on Treatment Platelet Reactivity and Genotype Variation: High Clopidogrel Dose Versus Prasugrel RESET GENE Trial
Brief Title: Therapy With High Clopidogrel Dose or Prasugrel Standard Dose Reduces the Platelet Reactivity in Patients With Genotype Variation RESET GENE Trial
Acronym: RESET GENE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gennaro Sardella (Other)
Responsible Party: Sponsor-Investigator, Gennaro Sardella, Associate Professor in Cardiology, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RESET GENE
Record Dates: First submitted 2011-10-28; First posted 2011-11-07 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2011-11

CONDITIONS: Acute Coronary Syndrome
Keywords: antiplatelet effect; prasugrel; clopidogrel; ACS
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high clopidogrel dose (Active Comparator): Patients will be randomized to this arm to receive before high clopidogrel dose and after crossover they will receive standard dose of prasugrel
  Interventions: Drug: Clopidogrel; Drug: prasugrel
- prasugrel standard dose (No Intervention): Patients will be randomized to this arm to receive before standard dose of prasugrel and after crossover they will receive high clopidogrel dose.

INTERVENTIONS:
Drug: Clopidogrel — Patient will be randomized to this intervention will receive in the first time the high clopidogrel dose and after 14 days we will change their therapy with standard dose of prasugrel (crossover).
  Arms: high clopidogrel dose
Drug: prasugrel — Patient will be randomized to this intervention will receive in the first time the standard dose of prasugrel and after 14 days we will change their therapy with high dose of clopidogrel (crossover).
  Arms: high clopidogrel dose

SUMMARY:
Dual antiplatelet therapy with aspirin and Clopidogrel for at least one year is essential in patients following an acute coronary syndrome (ACS) or percutaneous coronary intervention (PCI) with drug eluting stent(s. Interindividual variability in platelet response to clopidogrel has been reported, with several mechanisms being implicated for high post-clopidogrel treatment PR. High on-treatment platelet reactivity (HTPR) is associated with an increased risk of adverse events after PCI. Studies in patients on chronic clopidogrel treatment are scarce, mainly in diabetic patients where HTPR is frequently present and independently predictive of adverse events. Optimization of platelet inhibition in patients with HTPR by increasing clopidogrel or alternatively, by more potent P2Y12 inhibitors is a controversial issue, mostly studied in post PCI patients, while no data exist, to the best of the investigators knowledge, in stable patients on chronic clopidogrel treatment. Therefore all HTPR patients, that will accept to participate, will be enrolled will randomize (Day 0) in a 1:1 ratio to either clopidogrel 150 mg a day, or prasugrel 10 mg a day, until Day 14 post randomization. A 14 ± 2 day visit will be performed for PR measurement and safety evaluation, with the blood sample being will be obtained 16-18 hours after the last study-drug dose, will follow by crossover directly to the alternate therapy for an additional 14 days without an intervening washout period. At Day 28 ± 2 patients will return for the clinical and laboratory assessment as did on Day 14 visit.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent to PCI
* lopidogrel resistance after Platelet reactivity blood test

Exclusion Criteria:

* history of bleeding diathesis
* chronic oral anticoagulation treatment
* contraindications to antiplatelet therapy
* PCI or coronary artery bypass grafting (CABG) <3 months
* hemodynamic instability
* platelet count <100,000/μl
* hematocrit <30%
* creatinine clearance <25 ml/min
* Patients with a history of stroke
* contraindication for prasugrel administration
* patients weighing <60 kg
* >75 years of age.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
antiplatelet effect of standard dose of prasugrel versus high dose clopidogrel in stable patients with HTPR | 14-28 days
  The primary aim will be to investigate the antiplatelet effect of standard dose of prasugrel versus high dose clopidogrel in stable patients with HTPR while receiving chronic clopidogrel treatment at the end of the 2 study periods (switching, crossover and post-crossover)

SECONDARY OUTCOMES:
Bleeding (major, minor, or minimal according to the TIMI study criteria) | 14-28 days
  Bleeding (major, minor, or minimal according to the TIMI study criteria)
Major Adverse Cardiac Cerebrovascular Events | 14-28 days
  cardiovascular death, myocardial infarction, and stroke

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Dept.of Cardiovascular Sciences,Policlinico Umberto I, Roma, Roma
  - Dept.of Cardiovascular Sciences,Policlinico Umberto I, Rome, Rome

REFERENCES:
- [Derived] Sardella G, Calcagno S, Mancone M, Palmirotta R, Lucisano L, Canali E, Stio RE, Pennacchi M, Di Roma A, Benedetti G, Guadagni F, Biondi-Zoccai G, Fedele F. Pharmacodynamic effect of switching therapy in patients with high on-treatment platelet reactivity and genotype variation with high clopidogrel Dose versus prasugrel: the RESET GENE trial. Circ Cardiovasc Interv. 2012 Oct;5(5):698-704. doi: 10.1161/CIRCINTERVENTIONS.112.972463. Epub 2012 Oct 9. PMID 23048056